CLINICAL TRIAL: NCT03675763
Title: Efficacy of a Craniosacral Therapy Protocol in the Treatment of Infant Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Mercedes Castejón Castejón, Osteopath, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77712133D
Record Dates: First submitted 2018-09-15; First posted 2018-09-18 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Infant Conditions; Colic, Infantile; Gastro-Intestinal Disorder
Keywords: Skull; Osteopathic Manipulation; Infantile Colic; Clinical Trial; Massage; Infant; Osteopathic Medicine
MeSH Terms: conditions — Colic; Digestive System Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Craniosacral therapy (Experimental): Craniosacral therapy and parent information on how to manage colic.
  Interventions: Other: Manual treatment
- Parent information (No Intervention): Parent information on how to manage colic.

INTERVENTIONS:
Other: Manual treatment — Craniosacral therapy protocol.
  Arms: Craniosacral therapy

SUMMARY:
This is a randomised controlled trial that aims to determine the effectiveness of craniosacral therapy for the treatment of infantile colic. Manual therapy was applied to a group of young infants diagnosed with colic while a second group did not received any treatment.

ELIGIBILITY:
Inclusion criteria:

* infants diagnosed with colic,
* with 0-90 days of age,
* who have had 3 hours of unexplainable crying per day for at least 3 days during the week previous to the study.

Exclusion criteria:

* infants diagnosed with any sort of pathological illness, allergies or food intolerance
* who have suffered any intracranial hemorrhages or skull fractures.

Ages: 0 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Crying | Change from baseline crying at 24 days, also evaluated at days 7 and 14
  Total amount of time the infant cries within a day. Crying is recorded by the parents in a diary. The higher the score is, the more hours of crying per day.

SECONDARY OUTCOMES:
Sleep | Change from baseline sleep at 24 days, also evaluated at days 7 and 14
  Total amount of time the infant sleeps within a day. Sleep is recorded by the parents in a diary. The higher the score is, the more hours of sleep per day.
Severity-ICSQ | Change from baseline severity -ICSQ at 24 days, also evaluated at days 7 and 14
  Severity of colic is measured according to a validated Infant Colic Severity Questionnaire. Minimum score is 24 and maximum 100. A score higher than 50 points suggests that the patient suffers from infantile colic.

IPD SHARING:
Plan to Share IPD: No